CLINICAL TRIAL: NCT01823952
Title: Phase 2, Single Centre, Randomized, Double-blind Study Conducted in Adult Males With Acute Dehydrating Diarrhea Due to Cholera With the Aim Being to Select One or More of the Three Fermentable Starches (FS) for an FS-HO-ORS Formulation.
Brief Title: High Amylose Maize Starch for Treatment of Cholera
Acronym: RESTORS
Status: Terminated | Type: Observational
Why Stopped: The study was closed early due to slow enrollment.
Sponsor: PATH (Other)
Responsible Party: Sponsor
Other Study IDs: RESTORS
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Diarrhea
Keywords: HAMS; ORS; Cholera; Diarrhea
MeSH Terms: conditions — Diarrhea; Cholera

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Analysis of the sample for starch, short chain fatty acids and faecal microbiota.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Males: Adult 18-65

SUMMARY:
A randomized, double-blind trial in adult males with acute dehydrating diarrhea of cholera comparing the safety, tolerability and efficacy of HAMS HO-ORS, HAMS 2.5% Acetate HO-ORS, HAMS 6% Acetate HO-ORS and HO-ORS.

The primary hypothesis is that at least one of the hypo-osmolar ORS containing high amylose maize starch 6% acetate (HAMSA6-HO-ORS), hypo-osmolar ORS containing high amylose maize starch 2.5% acetate (HAMSA2.5-HO-ORS) and a hypo-osmolar ORS containing high amylose maize starch (HAMS-HO-ORS), will significantly reduce diarrhea duration compared with hypo-osmolar (HO) ORS.

Specifically, the investigators expect that HAMSA6 will be the most effective preparation.

DETAILED DESCRIPTION:
* Burden: Watery diarrhea including cholera continues to be a major cause of childhood mortality in developing countries, with an estimated 1.5 million children dying each year. This figure has greatly reduced from approximately 5 million diarrheal deaths annually 20 years ago, a phenomenon often attributed to the utilization of oral rehydration solution (ORS).
* Knowledge Gap: ORS is very effective in correcting dehydration and reducing mortality, but is not adequately used in many countries, partly due to the fact that it does not reduce diarrhea. The physiological basis for ORS is that glucose-stimulated sodium and fluid absorption is not inhibited by cyclic 3',5'-adenosine monophosphate (cAMP) and other diarrhea mediators which inhibit sodium chloride absorption. The conventional glucose-based ORS does not reduce duration or severity of diarrhea and may in fact paradoxically increase fecal fluid losses. Advances in ORS composition have included the universal adoption of hypo-osmolar ORS (HO-ORS) in 2003. Recent technological innovations have led to the use of amylase-resistant starches and their modifications in the treatment of diarrhea. Short chain fatty acids (SCFA), which are produced in colon from these non-absorbed carbohydrates, enhance sodium absorption. An orally administered, non-absorbed starch (i.e., one resistant to digestion by amylase) significantly reduced fecal fluid loss and the duration of diarrhea in patients with cholera.
* Relevance: Efforts are continuing to improve the efficacy of oral rehydration solution. As glucose stimulates sodium and water absorption in small intestine, short chain fatty acids (SCFAs) stimulate sodium and water absorption in the colon. In cholera, colonic function is also impaired due to the lack of SCFAs. The main source of SCFAs is the unabsorbed carbohydrates that are fermented in the colon by the colonic bacteria. The maize starch contains substantial amount of amylase resistant starch that escapes digestion and absorption in the small intestine and is fermented in the colon, liberating SCFAs. We expect that our experimental ORS containing maize starch will reduce the severity (stool volume) and enhance recovery (reduce duration) of diarrhoea.

ELIGIBILITY:
INCLUSION CRITERIA:

A participant is considered eligible for participation in the trial if the following inclusion criteria are satisfied on admission (Day 1, before randomization) to the hospital:

1. Participant is a male between 18 and 65 years of age inclusive
2. Severe watery diarrhea without fecal blood of less than 48 hours (with passage of 3 or more watery stools in the 24 hours before admission)
3. Signs of severe dehydration as per ICDDR,B guidelines (modified WHO guideline)
4. Dipstick test/Dark-field examination positive for Vibrio cholera
5. Written informed consent is provided
6. Participant is willing and able to comply with all trial requirements

EXCLUSION CRITERIA:

A participant who meets any of the following criteria on admission (before randomization) to the hospital will not qualify for the study

1. Evidence or history of any clinically significant illness as per the Investigator's discretion.
2. Known case of HIV or Hepatitis B
3. History of cancer
4. Known renal disease
5. Frequent excessive alcohol use, binge drinking (e.g. men consume 5 or more drinks in about 2 hours) or use of illicit drugs within the past two years
6. History of receiving antimicrobial or anti-diarrheal medication (loperamide, diphenoxylate, etc.) within seven days of admission
7. Concomitant infection requiring antimicrobial therapy
8. Donated blood or plasma or experienced clinically significant loss of blood within eight weeks prior to admission or who plan to donate blood within 1 month after study participation
9. Clinically significant abnormal laboratory test results as determined by the investigator
10. Treatment within 30 days prior to admission (or five half-lives of the compound, if longer) with any investigational agent or device
11. History of seizure (including febrile seizure) or loss of consciousness;
12. History of any GI Surgery related to Bowel resections and gastric anastomoses in past except Appendicitis
13. For any reason, deemed by the investigator to be inappropriate for this study, including participants who are unable to communicate or to cooperate with the investigator or designee
14. Prior enrolment in this trial

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population is 150 adult male patients: 40 each in the HAMS, HAMSA2.5 and HAMSA6 arms and 30 in the HO-ORS study arm.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Duration of Diarrhea | 12 hrs w/o diarrhoea, up to max of 96 hrs
  Criteria evaluated:
  Duration of diarrhea during the study period (defined as time from randomisation to the last watery stool preceding two soft/formed stools or a 12 hour period without diarrhea, up to a maximum of 96 hours)

SECONDARY OUTCOMES:
Stool output and fluid intake rate | 0 to 96 hrs
  Criteria evaluated:
  * Total output of watery stool (g/kg body weight)
  * Weight of watery stool
  * Intake of oral fluids including ORS and plain water in mL/kg from time of randomization to the first soft/formed stool or 48 hours of treatment with study products, whichever is sooner
  * Proportion of patients who vomit in the first 24 hours
  * Proportion of patients who require unscheduled intravenous fluids post randomization
  * Amount (mL/kg) of unscheduled intravenous fluids required post randomization
  * Proportion of patients with diarrhea beyond 48 hours

OTHER OUTCOMES:
Safety & Tolerability as measured by adverse events, vital signs and lab parameters | Approximately 24 hours after randomization
  * Proportion of patients with biochemical and symptomatic hyponatremia
  * Proportion of patients with adverse events deemed possibly or definitely related to treatment with the investigational products
  * Proportion of patients with abnormal biochemical and haematological values (any grade 3 as per CTCAE version IV criteria or above)
  * Proportion of patients with serious adverse events deemed possibly or definitely related to treatment with investigational products

CONTACTS AND LOCATIONS:
Overall Officials: Nur H Alam, MD MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital - icddr,b (International Centre for Diarrhoeal Disease Research, Bangladesh), Mohakhali, Dhaka Division, Bangladesh